CLINICAL TRIAL: NCT04689997
Title: Online System for Primary Care to Prevent and Address Teen Substance Use
Acronym: Substance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Total Child Health, Inc. (Industry)
Collaborators: Boston Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R44DA046262 (NIH)
Record Dates: First submitted 2020-12-25; First posted 2020-12-30 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Substance Use
Keywords: substance use
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: We will employ a cluster randomized two-group pretest-posttest design, clustered at the provider level.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participating teens and parents will not know that their primary care provider has extra tools for their health supervision visit devoted to substance use prevention, reduction, or care. Statisticians will be blind to assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- computerized Substance Brief Intervention cSBI (Experimental): Enhanced care PCPs will address the serious morbidity of teen substance use during routine check-up visits using cSBI and follow up care using a new Module of CHADIS that facilitates guideline-based care. The CHADIS c-SBI Module will include pre-visit screening tools and embedded education that cover substance use and strengths and goals. It will also include reminders to the patient about their goals and commitments for change and teleprompted interview hints for the PCP. These hints will be aimed at enhancing a patient focused discussion of individual strengths and barriers related to the teens' goals in a motivational interviewing style.
  Interventions: Behavioral: cSBI
- Standard care (No Intervention): Standard care PCPs will screen using a standard SU tool and carry out their usual health supervision visits without additional decision support.

INTERVENTIONS:
Behavioral: cSBI — The standard CRAFFT SU screen has additional questions about reasons to use or not use, SU expectancies of effect and embedded education. The teens of enhanced care PCPs will also complete a Strengths and Goals tool. Data from both will be used by the PCP in counseling regarding continued abstention, reduction or cessation of SU or referral. Teens will also get monthly text messages about goals.
  Arms: computerized Substance Brief Intervention cSBI

SUMMARY:
This Quality Improvement (QI) project for physician education will build on an existing platform, CHADIS (Comprehensive Health and Decision Information System; www.CHADIS.com). We plan to further develop and test innovations that will assist primary care providers (PCPs) in addressing the serious morbidity of teen substance use during routine check-up visits and follow up care using a new Module of CHADIS that facilitates guideline-based care. The CHADIS c-SBI (computer-facilitated Substance screening and provider Brief Intervention) Module will include pre-visit screening tools that cover substance use and strengths and goals. It will also include reminders to the patient about their goals and commitments for change and a teleprompter for interview hints for the PCP. These hints will be aimed at enhancing a patient focused discussion of individual strengths and barriers related to the teens' goals in a motivational interviewing style.

DETAILED DESCRIPTION:
The primary goals of this project are to develop and test an innovative teen substance use (SU) module in CHADIS integrating the cSBI questionnaire and decision support into CHADIS along with teen strength and goal data to be called CHADIS-cSBI. The CHADIS-cSBI will facilitate evidence-based SU screening, severity assessment and initiation of primary care management and care coordination for any referrals to reduce morbidity, mortality and costs of SU. Inclusion of strength and goal data is anticipated to foster the doctor-teen relationship and make SU advice more effective.

Primary Research Questions

1. Of those who reported any substance use at their annual well-visit, is there a lower rate of reported use at 3- and 12- months follow-up among those exposed to CHADIS-cSBI as compared to those who received treatment as usual?
2. Of those who reported no substance use at their annual well-visit, is there a lower rate of reported use at 3- and 12- months follow-up among those exposed to CHADIS-cSBI as compared to those who received treatment as usual? Secondary Research Question

1) Among all patients, is there are lower rate of reported driving after using or riding with a driver who has been using substances (risky driving/riding) at 3- and 12-months follow-up among those exposed to CHADIS-cSBI as compared to those who received treatment as usual? We will employ a cluster randomized two-group pre-test-post-test design, clustered at the provider level. Given the nature of the enhanced care and the measurement it is not possible to randomize at the patient level, and it is not necessary to randomize at the clinic level. The use of a cluster-randomized design adds complexity, and generally requires larger samples to achieve sufficient statistical power as compared to simple randomized control trials. Sample size estimates consider the design effect resulting from a cluster randomized design as well as other assumptions.

A total of 40 PCPs reporting at least 2 teen well visits per week, either in person or by telemedicine visit, will be recruited and randomly assigned in equal numbers to the enhanced care and standard care arms of the study. We will randomize clinicians stratified by whether they have completed Adolescent Medicine fellowships, as those with Adolescent Medicine training have been shown to have higher rates of addressing substance use in their practice. The authors' prior experience showed that, in a trial where the patients were randomized, individual PCPs being trained to deliver the counseling did not give similar levels of counseling to intervention and control patients. Their studies also show wide variation in patient-reported receipt of counseling across participating providers; e.g., within the intervention group, there was a range from 65%-93% across providers within one site. Such heterogeneity within a site reduces concern about contamination of practice across providers. All 12-18 year old patients in the practice will complete pre-visit screens dependent on the randomization of their own attributed PCP. While there are, in fact, three levels (i.e., patient -> practitioner -> practice), we confine the fundamental design herein to two levels (i.e., patient -> practitioner). Intra-class correlations will be used to adjust sample size estimates during power analyses, and also used to account for the covariance that is presumed to exist wherein patients from the same cluster (i.e., PCP) are likely to be more similar to each other than to patients from other clusters. The study design is depicted by the following research design notation figure:

T0 T1 T2 T3 NR O X O O NR O O O

Each line represents the study timeline for an enhanced care group (i.e., first line represents the CHADIS-cSBI group; second line represents the Standard CHADIS group using CRAFFT), N: Indicates the groups are nonequivalent (i.e., subjects are not randomly assigned to treatment).

R: Indicates the groups are derived from randomly assigned PCPs (i.e., the subjects are treated by clinicians randomly assigned to a treatment protocol).

O: Indicates an observation timepoint (i.e., data collection). The first observation (T0) represents baseline substance use for patients at their well-visit; the second and third refer to follow-up assessments at 3 and 12 months post-visit.

X: Indicates the enhanced care (i.e., CHADIS-cSBI) that patients of enhanced care providers will receive.

Finally, because this will be a Quality Improvement study, and practical utility of the CHADIS-cSBI enhanced care applies at the practitioner level rather than the patient level, we will conduct all analyses using Intent to Treat groups, retaining all patients initially enrolled regardless of participation or compliance.

ELIGIBILITY:
Inclusion Criteria:

* English speaking and reading

Exclusion Criteria:

* None

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 5000 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Substance use level | Change from Day 0 to 3 months
  Repeated CRAFFT screens at 3 months documenting SU level.
Substance use at one year | Change from Day 0 to 11.5 months
  Repeated CRAFFT screens at 3 months documenting SU level.

SECONDARY OUTCOMES:
Riding/driving risky behavior | Change from Day 0 to 3 months
  rate of reported driving after using or riding with a driver who has been using substances
Riding/driving risky behavior | Change from Day 0 to 11.5 months
  rate of reported driving after using or riding with a driver who has been using substances

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J Howard, MD, Principal Investigator — CHADIS aka Total Child Health; Raymond Sturner, MD, Principal Investigator — Center for Promotion of Child Devlopment; Sion Harris, PhD, Principal Investigator — Boston Children's Hospital; Lydia Shrier, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Total Child Health dba CHADIS, Inc., Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Only group deidentified data will be shared to qualified researchers after the study results have been reported.